CLINICAL TRIAL: NCT02707172
Title: Soap and the Removal of Diethylhexyl Phthalate From Hands: N-of-1 and Cross-Over Designs
Brief Title: Removal of Dermal Exposure to Phthalate Ester by Hand Washing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Principal Investigator, Ming-Tsang Wu, Director of Center of Environmental & Occupational Medicine, Kaohsiung Medical University Chung-Ho Memorial Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: KMU-PH-201301
Record Dates: First submitted 2016-03-03; First posted 2016-03-14 (Estimated); Results first posted 2017-04-14 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-09

CONDITIONS: Environmental Exposure; Exposure to Pollution
Keywords: Diethylhexyl Phthalate; Hand hygiene; Soaps; N-of-1 design; Cross-Over Studies
MeSH Terms: interventions — Hand Disinfection; Soaps; Water

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Subject was first exposed to 1000 microgram of diethylhexyl phthalate on both hands, and was asked to perform the intervention, handwashing with soap, by a standardized hand washing technique.
  Then the subjects in this arms are crossover to receive placebo, handwashing with water only.
  Interventions: Behavioral: handwashing with soap; Behavioral: handwashing with water
- Placebo (Placebo Comparator): Subject was exposed to 1000 microgram of diethylhexyl phthalate on both hands, and was asked to perform the placebo, handwashing with water, by a standardized hand washing technique.
  Then the subjects in this arms are crossover to perform the intervention, handwashing with soap.
  Interventions: Behavioral: handwashing with soap; Behavioral: handwashing with water

INTERVENTIONS:
Behavioral: handwashing with soap — handwashing with soap by a standardized 6-step handwashing technique
Behavioral: handwashing with water — handwashing with water by a standardized 6-step handwashing technique

SUMMARY:
The aim of the study is to evaluate the effectiveness in removing chemical exposure on hand, the investigators compare removal efficiency of Di-(2-ethylhexyl)phthalate (DEHP) on hands by hand washing with soap and water vs. water only. In two three-day N-of-1 trials, residual DEHP was measured in a single female adult who washed exposed hands with soap-and-water or water-only. Subsequently, a crossover study was performed by randomly assigning another 28 subjects equally to wash with soap-and-water or with water-only, and then each one received the other treatment 24 hrs later.

DETAILED DESCRIPTION:
Three studies, consisting of two N-of-1 trials and one crossover study, were used to compare the effect of handwashing with soap and water (intervention) and handwashing with water only (placebo) on phthalate removal from hands. The soap was plain soap, consisting of vegetable oil and sodium hydroxide. First, the investigators recruited one healthy female aged 25 yrs to participate in two N-of-1 trials. In each trial, her hands would be exposed to DEHP and then be treated with either soap intervention or placebo for three times over the course of three days. The first trial started on 15 May 2013. On day one, after the subject prewashed her hands, she allowed her hands to be exposed to a designated amount of DEHP. She then washed them with water only and rinsed them sequentially in three separate polyethylene (PE) bags, each containing 200 mL water to collect DEHP residue. One hour later, the same protocol was followed, except the exposed hands were treated with soap and water instead of water only (Figure 1a). The water rinsing in three separate bags remained the same. The pairs of studies were repeated on two subsequent days (16 and 17 May).

In the second N-of-1 trial, which was also performed over three days (22-24 May), the protocol using the same subject remained the same for all three days, except that the subject underwent intervention first then placebo. The water rinsing remained the same.

A randomized 2 × 2 crossover study was subsequently conducted between June and September 2013. The investigators assigned one group of 7 females and 7 males to perform handwashing with soap and water (intervention) and another group of 7 females and 7 males to perform handwashing with water only (placebo). Briefly, on the first day, the two groups washed their DEHP exposed hands using either soap and water or water only and then rinsed them in a PE bag with 200 mL water to collect DEHP. After 24 hrs, the experiment was crossed-over with the same two groups receiving the opposite treatments.

ELIGIBILITY:
Inclusion Criteria:

* healthy adult over age of 18 years
* BMI>18

Exclusion Criteria:

* diagnosis of any type of cancers, dermatitis, asthma
* cut, abrasion, and trauma on hands
* BMI <18

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-05; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Tsang Wu, ScD, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University, Kaohsiung City, Kaohsiung County, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Kaohsiung Medical university in Kaohsiung City, Taiwan from May, 2013 to September, 2013.
Groups:
- All Participants: All participants underwent two experiments, one with placebo (handwashing with water) and one with intervention (handwashing with soap), but in different order.
  28 participants underwent placebo first and crossed-over to received intervention; while the other 28 participants underwent intervention first and then placebo. There was one day wash-out period between the two sets of experiment.
  In each set of the experiment, each participant was exposed to 1000 microgram of diethylhexyl phthalate on both hands, and was asked to perform the placebo or intervention by a standardized hand washing technique depending on the sequence assignment.
  A total of 56 placebo experiments were performed and a total of 56 intervention experiments were performed in the study.
Period: 1st Set of Experiment
Arm/Group | All Participants
Started | 28
Completed | 28
Not Completed | 0
Period: Wash Out
Arm/Group | All Participants
Started | 28
Completed | 28
Not Completed | 0
Period: 2nd Set of Experiment
Arm/Group | All Participants
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: A total of 28 participants were recruited and were divided into two groups, one group receiving placebo first and then intervention, the other group receiving intervention first and then placebo.
  The placebo is handwashing with water using the 6-step standardized handwashing technique.
  The intervention is handwasahing with soap using the 6-step standardized handwashing technique.
Arm/Group | All Participants
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.9 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 14
Region of Enrollment [Number; unit: participants]
  Taiwan | 28

OUTCOME MEASURES:

1. Primary Outcome: Amount of Diethylhexyl Phthalate Removed From Hand
Description: Water rinse were performed immediately after hand-washing, and the concentration of diethylhexyl phthalate in the soiled water is measured.
Time Frame: immediately right after hand-washing
Population: Each participant underwent two sets of experiments, one with placebo and one with intervention. 14 participants received placebo first and were crossed-over to received intervention. The other 14 participants received intervention first and were crossed-over to received placebo.
Measure: Mean (Standard Deviation); unit: percentage of DEHP removed
Arm/Group | All Participants
Number analyzed (Participants) | 28
percentage of DEHP removed
  Intervention | 94.64 (6.49)
  Placebo | 8.74 (5.69)

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Intervention: Subject was first exposed to 1000 microgram of diethylhexyl phthalate on both hands, and was asked to perform the intervention, handwashing with soap, by a standardized hand washing technique.
  Then the subjects in this arms are crossover to receive placebo, handwashing with water only.
  handwashing with soap: handwashing with soap by a standardized 6-step handwashing technique
  handwashing with water: handwashing with water by a standardized 6-step handwashing technique
- Placebo: Subject was exposed to 1000 microgram of diethylhexyl phthalate on both hands, and was asked to perform the placebo, handwashing with water, by a standardized hand washing technique.
  Then the subjects in this arms are crossover to perform the intervention, handwashing with soap.
  handwashing with soap: handwashing with soap by a standardized 6-step handwashing technique
  handwashing with water: handwashing with water by a standardized 6-step handwashing technique
Arm/Group | Intervention | Placebo
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No